CLINICAL TRIAL: NCT02776956
Title: Study on Left Atrial Function of Atrial Fibrillation After Radiofrequency Ablation With Statin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xieruiqin (Other)
Responsible Party: Sponsor-Investigator, xieruiqin, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xierqdoctormd
Record Dates: First submitted 2016-04-29; First posted 2016-05-19 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation;left atrial function
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- atorvastatin group (Experimental): atrial fibrillation in atorvastatin group will orally receive atorvastatin before and after operation.
  Interventions: Drug: atorvastatin group
- non-atorvastatin group (Other): atrial fibrillation in non-atorvastatin group will not receive atorvastatin before and after operation..
  Interventions: Drug: non-atorvastatin group

INTERVENTIONS:
Drug: atorvastatin group — Patients in atorvastatin group will orally receive 20 mg of atorvastatin per night (Pfizer) for three days before the operation and three months after the operation
  Arms: atorvastatin group
Drug: non-atorvastatin group — Patients in non-atorvastatin group will not receive atorvastatin before the operation and after the operation.
  Arms: non-atorvastatin group

SUMMARY:
A total of 120 patients with persistent atrial fibrillation (including continuous and long-standing persistent atrial fibrillation) and 60 patients with paroxysmal atrial fibrillation will receive radiofrequency ablation. Patients in each group will be randomly allocated into the statin treatment group and non-statin treatment group (allocation ratio, 1:1). Left atrial appendage flow velocity of all patients are measured by Transesophageal Echocardiography(TEE) 24 hours before the operation. Real-time ultrasound examinations of left atrial function are carried out for all patients before the operation and after the operation. Blood samples are extracted in all patients before the operation and after the operation. This study will clarify whether the application of statin drugs can improve postoperative left atrial function. This study will identify the time course and influence factors of left atrial recovery of atrial fibrillation after the operation to guide the time and the degree of anticoagulation and effectively prevent thromboembolic events. At the same time, biochemical indicators are detected to analyze which indicators are related to the postoperative recurrence of atrial fibrillation, the incidence of postoperative thrombosis and the recovery of postoperative left atrial function. Furthermore, this study will investigate whether the application of statin drugs can improve postoperative left atrial function by affecting these indicators.

ELIGIBILITY:
Inclusion Criteria:

* All persistent or permanent AF patients with refractory or intolerant to at least one Class 1 or Class 3 antiarrhythmic medication.
* paroxysmal atrial fibrillation with refractory or intolerant to at least one Class 1 or Class 3 antiarrhythmic medication.
* age is <80 years

Exclusion Criteria:

* left ventricular dysfunction
* LA >50 mm
* atrial thrombosis
* valvular heart disease
* hyperthyroidism
* patients who underwent prosthetic heart valve replacement
* patients with previous history of atrial fibrillation ablation
* Hyperlipidemia
* pregnant women
* patients with existing liver and kidney disease
* malignant tumors
* hematological system diseases

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-04; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Left atrial function of postoperative atrial fibrillation detected | 1-12 month

SECONDARY OUTCOMES:
Plasma biomarkers of inflammation,myocardial injury and prothrombotic assessed | 1-3 month

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China